CLINICAL TRIAL: NCT06884462
Title: Effect of High-intensity Laser Exercise Versus Moderate-intensity Aerobic Exercise on Diabetic Polyneuropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: physio 1 2025
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIL treatment group (Experimental): 30 patients with DPN who were advised to undergo HIL treatment for eight weeks
  Interventions: Radiation: High-intensity laser (HIL)
- Moderate-intensity aerobic exercise group (Experimental): 30 patients receive moderate-intensity aerobic exercise
  Interventions: Procedure: moderate-intensity aerobic exercise

INTERVENTIONS:
Radiation: High-intensity laser (HIL) — The wavelength measured 1064 nm, accompanied by a power output of 5.00 W. The frequency employed was 25 Hz
  Arms: HIL treatment group
Procedure: moderate-intensity aerobic exercise — walking on a treadmill at a speed of 3-4 miles per hour on a flat surface (0% incline) for 40 minutes, 3 times weekly over eight weeks
  Arms: Moderate-intensity aerobic exercise group

SUMMARY:
Diabetic poly neuropathy (DPN) is a length-dependent, symmetrical sensorimotor poly neuropathy and is among the most prevalent and challenging consequences of diabetes4.

The documented prevalence of DPN varies between 13% and 55%, with 25% to 50% of these individuals experiencing neuropathic pain5. This study was conducted to find out the impact of high-intensity laser versus moderate-intensity aerobic exercises on diabetic poly neuropathy patients.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic symptoms in the lower limbs, including numbness, tingling, pain, burning, electric shock, and stabbing

Exclusion Criteria:

* sensory polyneuropathy unrelated to diabetes as
* systemic diseases,
* infections,
* inflammatory conditions,
* drug effects,
* metal exposure,
* hereditary factors

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Lower extremity functional performance | 3 months
  scale for both groups from 0 (minimum) to 80 (maximum)

CONTACTS AND LOCATIONS:
Locations (1):
- Soad, Minya, Egypt